CLINICAL TRIAL: NCT02864147
Title: Treatment of High-Grade Pre-Neoplastic Cervical Lesions (CIN 2/3) Using a Novel "Prime and Pull" Strategy
Brief Title: Treatment of High-Grade Pre-Neoplastic Cervical Lesions (CIN 2/3)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1603017415; 000 (Other: YCTGT)
Record Dates: First submitted 2016-08-04; First posted 2016-08-11 (Estimated); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervical Dysplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Imiquimod

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- imiquimod + 9-valent HPV vaccine (Experimental): Participants randomized to the imiquimod + 9-valent HPV vaccine group will receive instruction on imiquimod self application (16 week course) at the baseline visit. In addition, all women (regardless of age) will be administered a dose of the HPV vaccine on day of enrollment (regardless of previous HPV vaccination history). Women previously unvaccinated will receive an additional booster dose at 8 weeks.
  Interventions: Drug: 9-valent HPV vaccine; Drug: Imiquimod
- imiquimod only (Active Comparator): Participants randomized to the imiquimod only group will receive instruction on imiquimod self application (16 week course) at the baseline visit.
  Interventions: Drug: Imiquimod
- observation only (control) (No Intervention): Participants randomized to the control group will only be observed and will receive no intervention.

INTERVENTIONS:
Drug: 9-valent HPV vaccine — All women (regardless of age) will be administered a dose of the HPV vaccine on day of enrollment (regardless of previous HPV vaccination history). Women previously unvaccinated will receive an additional booster dose at 8 weeks.
  Arms: imiquimod + 9-valent HPV vaccine
Drug: Imiquimod — At the baseline visit, this group will be instructed about the correct method of self-application of imiquimod 6.25mg as a vaginal suppository and receive a 16 week course of the drug.
  Arms: imiquimod + 9-valent HPV vaccine; imiquimod only

SUMMARY:
This is a randomized Phase II, three arm control trial in patients with Cervical Intraepithelial Neoplasia (CIN) 2/3 high grade cervical dysplasia. Patients with CIN 2/3 meeting eligibility criteria will have cervical biopsy specimens centrally reviewed by study pathologist to confirm diagnosis. HPV DNA test and HPV 16/18 genotyping will be performed from endocervical cytobrush samples to determine HPV status associated with the dysplasia.

Patients who have CIN 2/3 with HPV+ disease will be enrolled in this study. Patients will be randomized to one of three arms: observation only (control), imiquimod only, imiquimod + 9-valent HPV vaccine.

DETAILED DESCRIPTION:
The primary objectives of this study are as follows:

* To determine treatment efficacy defined as histologic regression to CIN 1 or less at weeks 20-24 (4 to 8 weeks after the end of imiquimod treatment) in the HPV Vaccine + Imiquimod group compared to control,
* To determine treatment efficacy defined as histologic regression to CIN 1 or less at weeks 20-24 (4 to 8 weeks after the end of imiquimod treatment) in the Imiquimod group compared to control.

The secondary objectives of this study are as follows:

* To assess complete regression (i.e., histologic remission) at weeks 20-24 (4 to 8 weeks after the end of imiquimod treatment) in each group,
* To assess HPV clearance in each group,
* To assess treatment tolerability.

In addition to the primary and secondary objectives of this study, there additional exploratory/correlative objectives. The exploratory/correlative objectives are as follows:

* To assess T cell infiltration in post-treatment cervical biopsies and endocervical cytobrush samples,
* To assess HPV16 E7 immunity in CD4/CD8 T cells.

ELIGIBILITY:
Inclusion Criteria

* Patients must have untreated cervical biopsy-proven, CIN 2/3 ectocervical lesion(s).
* Patients must have satisfactory colposcopy with visualization of the entire transformation zone or a negative endocervical curettage if colposcopy is unsatisfactory.
* Patients must be high-risk HPV+ as determined by commercially available DNA hybridization test which tests for 13 high-risk HPV types.
* All Patients must have a histologic diagnosis of CIN 2,3 cervical lesion(s) confirmed by a study pathologist within past 10 weeks.
* Patients must have signed an approved informed consent.
* Patients of childbearing potential must have a negative urine pregnancy test within 7 days prior to the study entry and be practicing an effective form of contraception.
* Patients must be at least 18 years of age based on previous and current cervical cancer screening guidelines.
* Patients must be fluent in speaking English or Spanish.

Exclusion Criteria

* Patients with unsatisfactory colposcopy* (unable to visualize entire transformation zone) or evidence of endocervical disease defined as CIN 2/3 diagnosed on endocervical curettage.

  *Patients with unsatisfactory colposcopy but negative endocervical curettage are eligible
* Patients with a history of invasive cervical cancer
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancers are excluded if there is any evidence of other malignancy being present within the last five years. Patients are also excluded if their previous cancer treatment contraindicates this protocol therapy.
* Patients with any unstable medical issue (including cardiac issues as above, active treatment for pulmonary embolism, CVA, renal or hepatic insufficiency, active infection/sepsis requiring IV antibiotics).
* Patients who have an uncontrolled seizure disorder, or active neurological disease.
* Patients known to be seropositive for HIV and active hepatitis, even if liver function studies are in the normal range. Patients otherwise immunocompromised will also be excluded (chronic steroid use, taking immunosuppressive medications).
* Pregnant or breastfeeding patients.
* Patients who have had a total hysterectomy (removal of uterus and cervix) or trachelectomy (removal of cervix).
* Patients with a known hypersensitivity to imiquimod. Patients with a known hypersensitivity to any prophylactic HPV vaccine or severe allergic reactions yeast (vaccine component).
* Patients who have received their first dose of HPV vaccine < 4 weeks ago or their second dose < 12 weeks ago.
* Known hypersensitivity or prior intravaginal treatment with Imiquimod

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2016-07; Primary Completion 2022-05-24 (Actual); Study Completion 2022-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro D Santin, MD, Principal Investigator — Yale University School of Medicine Department of Obstetrics, Gynecology & Reproductive Sciences, Division of Gynecologic Oncology; Sangini S Sheth, MD, MPH, Principal Investigator — Yale University School of Medicine Department of Obstetrics, Gynecology & Reproductive Sciences, Division of Gynecologic Specialties
Locations (1):
- Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Observation Only (Control) | Imiquimod Only | Imiquimod + 9-valent HPV Vaccine
Started | 45 | 45 | 43
Completed Treatment | 45 | 45 | 43
Placed On Follow Up | 29 | 35 | 28
Completed | 38 | 38 | 38
Not Completed | 7 | 7 | 5
Not completed — Withdrawal by Subject | 3 | 2 | 1
Not completed — Lost to Follow-up | 0 | 4 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Pregnancy | 4 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Opted for excisional procedures | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Observation Only (Control) | Imiquimod Only | Imiquimod + 9-valent HPV Vaccine | Total
Number analyzed (Participants) | 45 | 45 | 43 | 133
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 45 | 45 | 43 | 133
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 45 | 43 | 133
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 5 | 5 | 19
  Not Hispanic or Latino | 35 | 36 | 38 | 109
  Unknown or Not Reported | 1 | 4 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 3 | 2 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 8 | 4 | 16
  White | 33 | 28 | 34 | 95
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 6 | 1 | 12
Region of Enrollment [Number; unit: participants]
  United States | 45 | 45 | 43 | 133

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Objective Response
Description: The major parameters of objective response to be assessed include treatment efficacy defined as histologic regression of cervical dysplasia to CIN 1 or less after the end of imiquimod treatment, HPV clearance and treatment tolerance. Objective response will be categorized as 'yes' or 'no' and included in the evaluations are the following criteria:
  * Histologic regression (HR): Histologic regression of all index lesions to CIN 1 or less after end of imiquimod treatment period.
  * Histologic remission (HM): Complete regression of cervical dysplasia at all index biopsy sites after end of imiquimod treatment period.
  * Persistent Disease (PR): One or more index lesions persists with CIN 2,3 high grade dysplasia or new lesions are identified colposcopically and histologically confirmed to be CIN 2,3.
  * Progressive Disease (PD): Worsening histology of an index lesion.
Time Frame: Between weeks 20 and 24 (approximately week 22)
Population: Complete case analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Imiquimod + 9-valent HPV Vaccine | Imiquimod Only | Observation Only (Control)
Number analyzed (Participants) | 38 | 38 | 38
Participants
  Histologic regression (HR) | 32 | 36 | 30
  Histologic remission (HM) | 0 | 0 | 0
  Persistent Disease (PR) | 6 | 2 | 8
  Progressive Disease (PD) | 0 | 0 | 0
Statistical Analysis 1: Comparison: Imiquimod Only vs Observation Only (Control); Test type: Superiority; p = 0.043, Fisher Exact — Control is used as the referent using one-sided Fisher's exact tests with a multiple comparison-adjusted p<0.025 significance level
Statistical Analysis 2: Comparison: Imiquimod + 9-valent HPV Vaccine vs Observation Only (Control); Test type: Superiority; p = 0.384, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Incidence of HPV Clearance
Description: HPV Clearance will be categorized as 'yes' or 'no' and the evaluations are the following criteria: HPV clearance will be measured by both the Roche cobas HPV Test utilized by pathology concomitant with the pap test at final study visit which assesses for presence of 14 high risk HPV types as well as HPV 16/18 genotyping performed by Santin Lab.
Time Frame: Between weeks 20 and 24 (approximately week 22)
Population: Complete case analysis- 2 participants in imiquimod + 9-valent HPV vaccine were not assessed at follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Imiquimod + 9-valent HPV Vaccine | Imiquimod Only | Observation Only (Control)
Number analyzed (Participants) | 36 | 38 | 38
Participants
  HPV Negative | 18 | 24 | 19
  HPV Positive | 18 | 14 | 19
Statistical Analysis 1: Comparison: Imiquimod Only vs Observation Only (Control); Test type: Superiority; p = 0.177, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Imiquimod + 9-valent HPV Vaccine vs Observation Only (Control); Test type: Superiority; p = 0.592, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to 24 weeks
Arm/Group | Observation Only (Control) | Imiquimod Only | Imiquimod + 9-valent HPV Vaccine
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45 | 1/43
Other Adverse Events (participants affected / at risk) | 5/45 | 38/45 | 36/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observation Only (Control) (N=45) | Imiquimod Only (N=45) | Imiquimod + 9-valent HPV Vaccine (N=43)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observation Only (Control) (N=45) | Imiquimod Only (N=45) | Imiquimod + 9-valent HPV Vaccine (N=43)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Congenital, familial and genetic disorders - Other, specify (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 3 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 3 (3) | 0 (0)
Fatigue (General disorders) | 0 (0) | 8 (8) | 7 (7)
Fever (General disorders) | 0 (0) | 5 (5) | 5 (6)
Flu like symptoms (General disorders) | 0 (0) | 21 (24) | 18 (20)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 2 (4) | 3 (3)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (2) | 2 (2)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 12 (14) | 7 (9)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (3)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1) | 18 (23) | 21 (27)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 4 (4) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 3 (4) | 3 (3)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 9 (13) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 1 (2)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-24): https://cdn.clinicaltrials.gov/large-docs/47/NCT02864147/Prot_SAP_000.pdf